CLINICAL TRIAL: NCT06028035
Title: A Pilot Study of Hemp Hull WFI (BB01) to Reduce Intestinal Permeability in IBS-Diarrhea With Evidence of Bile Acid Diarrhea
Brief Title: A Study of Hemp Hull WFI for IBS Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-005827
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-10

CONDITIONS: Irritable Bowel Syndrome-bile Acid Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BB01 Supplement Bars (Experimental): Subjects will consume two BB01 supplement bars daily for 21 days.
  Interventions: Dietary Supplement: BB01

INTERVENTIONS:
Dietary Supplement: BB01 — 20 grams minimally processed form of Hemp hulls in the form of a bar/wafer.

SUMMARY:
The purpose of this study is the effect of a study bar, which contains 15 grams of insoluble dietary fiber total sourced from Hemp hulls, on intestinal permeability in irritable bowel syndrome (IBS)-bile acid diarrhea individuals.

DETAILED DESCRIPTION:
Patients with irritable bowel syndrome-bile acid diarrhea (IBS-BAD) have no evidence of significant histologically-evident inflammation or ulceration. The condition is often unrecognized in comparison with natural variations in bowel function in the general population. Hemp seeds are a complete source of protein, providing all nine essential amino acids, as well as polyunsaturated fats, especially omega-3 fatty acid, fiber, minerals and vitamins. Hemp hulls, the outer shell of the seeds, are typically rich in dietary fiber and phenolics and showed to have a beneficial effect on gut barrier function in vitro.

To demonstrate reduced intestinal permeability after 3 weeks of BB01 (20g of BB01, which reflects 15g of insoluble dietary fiber) consumption in a group of 10 patients with IBS-diarrhea with evidence of bile acid diarrhea, a group that has been previously documented to have increased GI permeability.

ELIGIBILITY:
Inclusion criteria

1. Prior diagnosis of bile acid diarrhea as documented by either

   1. total bile acid in 48 hour stool excretion of 2337 micromoles per 48 hours, or
   2. greater than 1000 micromoles per 48 hours with greater than 4% primary bile acids in stool, or
   3. greater than 10% primary bile acid (CA and CDCA) in stool 48 hour collection, or
   4. serum 7 alpha C4 greater than 52 ng/mL
2. BMI <40 kg/m2.
3. Prior cholecystectomy, appendectomy, and tubal ligation or hysterectomy will all be permissible for participation in the study.
4. Participants receiving bile acid sequestrant will not be permitted to continue therapy. and need to stop one week before baseline test.
5. No use of oral antibiotics and NSAIDs for 2 weeks prior to study treatment

Exclusion criteria

1. Diabetes mellitus (type 1)
2. Diabetes mellitus type 2 if taking metformin or GLP-1 agonist treatment (exenatide, liraglutide, semaglutide)
3. Uncontrolled hypertension (with BP measured >140/90mmHg in the CRTU)
4. BMI ≥40 kg/m2
5. Chronic NSAID use (>1 day/week)
6. Use of oral antibiotics and NSAIDs for 2 weeks prior to and during the entire 21 day study period
7. Use of bile acid sequestrant for 1 week prior to and during the entire 21 day study period
8. Diagnosis of gastrointestinal diseases that are associated with inflammation such as inflammatory bowel diseases and celiac disease or gastrointestinal infection in the prior 4 weeks;
9. Prior intestinal or colonic resection; note prior cholecystectomy, appendectomy, and tubal ligation or hysterectomy will all be permissible for participation in the study
10. Participation in highly vigorous exercise such as running >5 miles per day in week prior to the permeability test

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in urinary excretion of 13^C-mannitol | Baseline, 3 weeks
  Percent urinary excretion of 13^C-mannitol
Change in urinary excretion of lactulose | Baseline, 3 weeks
  Percent urinary excretion of lactulose

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No